CLINICAL TRIAL: NCT06035081
Title: CIRcadian Rhythms and CortisoL. Effects on Substrate Metabolism and Clock Gene Expression and Functioning
Acronym: CIRCLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1-10-72-83-22
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Healthy
Keywords: glucocorticoids; circadian rhythm; metabolism
MeSH Terms: interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prednisolone first, then placebo (Experimental): Prednisolone 12.5 mg twice daily for 5 days. Placebo twice daily for 5 days
  Interventions: Drug: Prednisolone; Other: Placebo
- Placebo first, then prednisolone (Experimental): Placebo twice daily for 5 days Prednisolone 12.5 mg twice daily for 5 days.
  Interventions: Drug: Prednisolone; Other: Placebo

INTERVENTIONS:
Drug: Prednisolone — see arm description
Other: Placebo — Placebo similar to prednisolone

SUMMARY:
The aim of this project is to study the effects of exogenous glucocorticoid exposure on substrate metabolism, energy expenditure and correlates of circadian rhythmicity in healthy adults. The hypotheses are:

Short-term high dose glucocorticoid exposure in healthy subjects disrupts:

* The inherent circadian pattern of the respiratory exchange ratio and REE
* Sleep quality, appetite and food intake
* Clock gene expression and function in adipose tissue, skeletal muscle and blood leukocytes

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* BMI 20-30 kg/m2
* Written informed consent

Exclusion Criteria:

* Any chronic disease requiring daily medication excluding atopic skin or hay fever
* Alcohol consumption >21 units per week
* Strong CYP3A4 inhibitors or inducers
* Use of glucocorticoid (GC) formulations: Inhaled corticosteroids, intra-articular or intramuscular injections, steroid creams European steroid group IV-V used in the genital area
* Permitted glucocorticoid formulations: eye-drops, nasal spray, GC creams European steroid group I-III, and European steroid group IV-V used in the non-genital area only
* Shift work
* Severe claustrophobia
* Use of melatonin
* Previous diagnosis of a sleep disorder
* Known severe sleep apnea (>30 respiration breaks/hour over 10 seconds)
* Deemed unable to complete the study safely by investigator

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-04-13 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Sleeping RER | Study day 1 and 2 (7 weeks apart)
  Change in respiratory exchange ratio (RER) during sleep between placebo and prednisolone
Change in TEE | Study day 1 and 2 (7 weeks apart)
  Change in Total Energy Expenditure between placebo and prednisolone
Change in REE | Study day 1 and 2 (7 weeks apart)
  Change in Resting Energy Expenditure between placebo and prednisolone and morning/evening
Change in RER from fasting to feeding | Study day 1 and 2 (7 weeks apart)
  Change in respiratory exchange ratio (RER) after standard meal between placebo and prednisolone and morning/evening

SECONDARY OUTCOMES:
Change in PAEE | Study day 1 and 2 (7 weeks apart)
  Change in Physical Activity related Energy Expenditure (PAEE) between placebo and prednisolone and morning/evening
Change in SEE | Study day 1 and 2 (7 weeks apart)
  Change in Sleeping Energy Expenditure (PAEE) between placebo and prednisolone
Change in DIT | Study day 1 and 2 (7 weeks apart)
  Change in diet-induced thermogenesis between placebo and prednisolone and prednisolone and morning/evening
Change in clock gene mRNA levels leukocytes | Study day 1 and 2 (7 weeks apart)
  Change in mRNA expression levels in blood leukocytes between placebo and prednisolone and prednisolone and morning/evening
Change in clock gene mRNA levels adipose tissue | Study day 1 and 2 (7 weeks apart)
  Change in mRNA expression levels in adipose tissue biopsies between placebo and prednisolone and prednisolone and morning/evening
Change in clock gene mRNA levels skeletal muscle | Study day 1 and 2 (7 weeks apart)
  Change in mRNA expression levels in skeletal muscle tissue biopsies between placebo and prednisolone and prednisolone and morning/evening
Change in appetite | Study day 1 and 2 (7 weeks apart)
  Measured by numerical rating scale on parameters hunger, fullness, satiety, desire and prospective consumption with values 1 (not at all) to 10 (maximally present) before and after ad libitum meal and standard meal, and between placebo and prednisolone and morning/evening. The scale is adapted from PMID: 20122136
Change in ad libitum food intake | Study day 1 and 2 (7 weeks apart)
  Measured by caloric intake between placebo and prednisolone and morning/evening
Change in food intake at home | Intervention period 1 and 2 (7 weeks apart)
  Measured by dietary registration during prednisolone and placebo
Change in fasting lipid oxidation rates | Study day 1 and 2 (7 weeks apart)
  Measured by whole room Indirect calorimetry between placebo and prednisolone and morning/evening
Change in lipid oxidation rates from fasting to fed | Study day 1 and 2 (7 weeks apart)
  Measured by whole room Indirect calorimetry between placebo and prednisolone and morning/evening
Change in glucose oxidation rates from fasting to fed | Study day 1 and 2 (7 weeks apart)
  Measured by whole room Indirect calorimetry between placebo and prednisolone and morning/evening
Change in fasting glucose oxidation rates | Study day 1 and 2 (7 weeks apart)
  Measured by whole room Indirect calorimetry between placebo and prednisolone and morning/evening
Change in fasting protein oxidation rates | Study day 1 and 2 (7 weeks apart)
  Measured by whole room Indirect calorimetry between placebo and prednisolone and morning/evening
Change in protein oxidation rates from fasting to fed | Study day 1 and 2 (7 weeks apart)
  Measured by whole room Indirect calorimetry between placebo and prednisolone and morning/evening
Change in ghrelin levels | Study day 1 and 2 (7 weeks apart)
  Measured in serum before and after ad libitum meals and standard meals; between placebo and prednisolone and morning/evening
Change in LEAP-2 levels | Study day 1 and 2 (7 weeks apart)
  Measured in serum before and after ad libitum meals and standard meals; between placebo and prednisolone and morning/evening
Change in GLP-1 levels | Study day 1 and 2 (7 weeks apart)
  Measured in serum before and after ad libitum meals and standard meals; between placebo and prednisolone and morning/evening
Change in GIP levels | Study day 1 and 2 (7 weeks apart)
  Measured in serum before and after ad libitum meals and standard meals; between placebo and prednisolone and morning/evening
Change in Glucose levels | Study day 1 and 2 (7 weeks apart)
  Measured in serum before and after ad libitum meals and standard meals; between placebo and prednisolone and morning/evening
Change in Insulin levels | Study day 1 and 2 (7 weeks apart)
  Measured in serum before and after ad libitum meals and standard meals; between placebo and prednisolone and morning/evening
Change in Glucagon levels | Study day 1 and 2 (7 weeks apart)
  Measured in serum before and after ad libitum meals and standard meals; between placebo and prednisolone and morning/evening
Change in Gastrin levels | Study day 1 and 2 (7 weeks apart)
  Measured in serum before and after ad libitum meals and standard meals; between placebo and prednisolone and morning/evening
Change in CCK levels | Study day 1 and 2 (7 weeks apart)
  Measured in serum before and after ad libitum meals and standard meals; between placebo and prednisolone and morning/evening
Change in cortisol levels | Study day 1 and 2 (7 weeks apart)
  Measured successively over 24 hours in serum during study days
Change in FAP cells in skeletal muscle | Study day 1 and 2 (7 weeks apart)
  Fibro-adipogenic progenitor cells levels and characteristics in skeletal muscle tissue biopsies between placebo and prednisolone and prednisolone and morning/evening
Change in FAP cells in adipose tissue | Study day 1 and 2 (7 weeks apart)
  Fibro-adipogenic progenitor cells levels and characteristics in adipose tissue biopsies between placebo and prednisolone and prednisolone and morning/evening
Change in physical activity levels | Intervention period 1 and 2 (7 weeks apart)
  Measured by actigraph during study periods
Change in IPAQ-7 | Intervention period 1 and 2 (7 weeks apart)
  Measured by Internation Physical Activity Questionnaire
Change in sleep quality (measured) | Intervention period 1 and 2 (7 weeks apart)
  Measured by actigraph during study periods
Change in sleep quality (reported) | Intervention period 1 and 2 (7 weeks apart)
  Measured by Pittsburgh Sleep Quality Index questionnaire
Change in sleep quality | Study day 1 and 2 (7 weeks apart)
  Measured by polysomnography
Change in HADS | Intervention period 1 and 2 (7 weeks apart)
  Measured by Hospital Anxiety and Depression Scale (HADS), a 14-question instrument with 7 questions measuring anxiety and 7 measuring depression. Each is scored between 0 (no impairment) and 3 (severe impairment)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Otto L Jørgensen, Professor, Study Director — Aarhus University Hospital; Simon B Hansen, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Endocrinology and Internal Medicine, Aarhus, State, Denmark

IPD SHARING:
Plan to Share IPD: No